CLINICAL TRIAL: NCT01402804
Title: Non-steroidal Anti-inflammatory Drugs Impair the Platelet Inhibiting Effect of Acetylsalicylic Acid in Coronary Artery Disease Patients
Brief Title: NSAIDs in Coronary Artery Disease Patients
Status: Completed | Type: Observational
Sponsor: Heinrich-Heine University, Duesseldorf (Other)
Responsible Party: Principal Investigator, Klinik für Kardiologie, Pneumologie und Angiologie, Klinik für Kardiologie, Pneumologie und Angiologie, Heinrich-Heine University, Duesseldorf
Other Study IDs: AGP-0001
Record Dates: First submitted 2011-07-25; First posted 2011-07-26 (Estimated); Last update posted 2013-11-11 (Estimated); Status verified 2013-11

CONDITIONS: CAD

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Stable CAD, ASA, NSAID
- Stable CAD, ASA

SUMMARY:
Introduction:

Different groups already showed in retrospective subgroup analyses, that there is an increased risk for cardiovascular events in patients on a simultaneous ASA/NSAID treatment.

Methods:

Light-Transmission aggregometry

Hypothesis:

Simultaneous administration of different NSAIDs and ASA impair the platelet inhibiting effect of ASA.

ELIGIBILITY:
Inclusion Criteria:

* Patients on a simultaneous ASA, NSAID treatment
* > 18 years

Exclusion Criteria:

* unconsciousness, not able to consent
* reanimation, cardiac shock

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with a stable CAD undergoing coronary angiography in the Universitätsklinik Düsseldorf.
Sampling Method: Non-Probability Sample
Enrollment: 85 (Actual)
Dates: Start 2011-07; Primary Completion 2013-07 (Actual); Study Completion 2013-07 (Actual)

PRIMARY OUTCOMES:
Thromboxane-levels and light-transmission aggregometry in response to arachidonic acid | During hospital stay

CONTACTS AND LOCATIONS:
Overall Officials: Amin Polzin, MD, Principal Investigator — Klinik für Kariologie, Pneumologie und Angiologie, Universtiätsklinikum Düsseldorf; Tobias Zeus, MD, Study Chair — Klinik für Kardiologie, Pneumologie und Angiologie; Thomas Hohlfeld, MD, Study Chair — Institut für Pharmakologie und Klinische Pharmakologie, Heinrich-Heine-Univerität Düsseldorf; Malte Kelm, MD, Study Director — Heinrich-Heine University, Duesseldorf
Locations (1):
- Heinrich-Heine-University, Düsseldorf, North Rhine-Westphalia, Germany

REFERENCES:
- [Derived] Achilles A, Mohring A, Dannenberg L, Piayda K, Levkau B, Hohlfeld T, Zeus T, Kelm M, Polzin A. Analgesic medication with dipyrone in patients with coronary artery disease: Relation to MACCE. Int J Cardiol. 2017 Jun 1;236:76-81. doi: 10.1016/j.ijcard.2017.02.122. Epub 2017 Feb 27. PMID 28262342
- See also: Related Info — http://www.uniklinik-duesseldorf.de/kardiologie